CLINICAL TRIAL: NCT04916509
Title: Treatment Patterns and Clinical Outcomes Among Patients Receiving Palbociclib Combinations for Hormone Receptor Positive (HR+)/Human Epidermal Growth Factor Receptor 2 Negative (HER2-) Advanced/Metastatic Breast Cancer in the Arabian Gulf Region Like Saudi Arabia, UAE and Other GCC Countries: A Retrospective Study (Treasure Study)
Brief Title: Treatment Patterns and Clinical Outcomes Among Patients Receiving Palbociclib Combinations for Hormone Receptor Positive (HR+)/Human Epidermal Growth Factor Receptor 2 Negative (HER2 ) Advanced/Metastatic Breast Cancer in the Arabian Gulf Region
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A5481136; TREASURE (Other: Alias Study Number)
Record Dates: First submitted 2021-05-19; First posted 2021-06-07 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Breast Neoplasms
Keywords: Retrospective Studies; palbociclib
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib; Fulvestrant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Palbociclib plus an aromatase inhibitor: Adult metastatic breast cancer patients who initiated Palbociclib + an aromatase inhibitor.
  Data will be retrospectively abstracted over an observational look-back period from 01st January 2015 to 30th September 2019.
  Aligned with Locally Approved Indication
  Interventions: Drug: Palbociclib plus an aromatase inhibitor
- palbociclib plus fulvestrant: Adult metastatic breast cancer patients who initiated Palbociclib + fulvestrant. Data will be retrospectively abstracted over an observational look-back period from 01st January 2015 to 30th September 2019.
  Aligned with Locally Approved Indication
  Interventions: Drug: Palbociclib plus fulvestrant

INTERVENTIONS:
Drug: Palbociclib plus an aromatase inhibitor — Palbociclib plus an aromatase inhibitor therapy
  Groups: Palbociclib plus an aromatase inhibitor
Drug: Palbociclib plus fulvestrant — Palbociclib plus fulvestrant
  Groups: palbociclib plus fulvestrant

SUMMARY:
retrospective non-interventional study (NIS) that aims to describe the demographics, clinical characteristics, clinical outcomes, and treatment patterns, among patients receiving palbociclib for the treatment of HR+/HER2- metastatic/locally advanced breast cancer (BC)

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old.
2. HR+/HER2- BC diagnosis with confirmed metastatic/locally advanced disease.
3. Patient initiated on palbociclib (regardless the line of therapy) within the period between 01st January 2015 and 01st March 2019.
4. Minimum of six months of follow up data since palbociclib initiation.
5. Received palbociclib plus aromatase inhibitor or palbociclib plus fulvestrant in line with the licensed indication(s).

Exclusion Criteria:

1. Prior or current enrolment in an interventional clinical trial for metastatic/locally advanced BC.
2. Patients who were initiated on palbociclib after 01st March 2019.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data will be abstracted from the medical records of all eligible patients across 17 - 35 selected sites from Arabian Gulf Region countries. The observational period for patients is the 57 month-period prior to the study index date. During this period, patients who initiated treatment with palbociclib between 01st January 2015 and 01st March 2019 will be considered eligible for participation in the study. Sites from diverse health care settings
Sampling Method: Probability Sample
Enrollment: 258 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2022-12-27 (Actual); Study Completion 2022-12-27 (Actual)

PRIMARY OUTCOMES:
Demographical Characteristics of Participants | Upon BC diagnosis up to date of index treatment (from data collected and observed retrospectively between 01 January 2015 and 01 March 2019)
Demographical Characteristics of Participants: Biomarker status | Upon BC diagnosis up to date of index treatment (from data collected and observed retrospectively between 01 January 2015 and 01 March 2019)
  Biomarker status - (estrogen receptor [ER], progesterone receptor [PR], HER-2 neu, Ki67, Germline BRCA [gBRCA] testing).
Clinical Characteristics of Participants: Description of diagnosis | Upon BC diagnosis up to date of index treatment (from data collected and observed retrospectively between 01 January 2015 and 01 March 2019)
  Description of diagnosis - staging, node status, menopause status, diagnosis for which palbociclib combination was prescribed, sites of metastases, de novo vs. recurrent disease.
Number of patients receiving adjuvant therapies | Upon diagnosis of BC (from data collected and observed retrospectively between 01 January 2015 and 01 March 2019)
  Adjuvant therapies received for the treatment of early or locally advanced breast cancer (Stages 0-IIIa) (if available)
Number of participants receiving treatment for advanced/metastatic BC before and after palbociclib combination use | Upon diagnosis of metastatic/locally advanced HR+/HER2 BC for a maximum of 4 years approximately (from data collected and observed retrospectively between 01 January 2015 and 01 March 2019)
  Treatments and supportive therapies received since metastatic/locally advanced HR+/HER2- diagnosis. Duration of treatments. Reasons for regimen changes. Starting dose, duration of treatment, changes in dose, interruptions, cycle delays and discontinuations. Where possible reasons for change in treatment. Line of treatment.
Number of participants with dose changes associated with palbociclib use | From 01 January 2015 to 30 September 2019
  Starting dose, duration of treatment, changes in dose, interruptions, cycle delays and discontinuations. Where possible, reasons for change in treatment. Line of treatment.
Number of participants to discontinue treatment associated with palbociclib use | From 01 January 2015 to 30 September 2019
  Starting dose, duration of treatment, changes in dose, interruptions, cycle delays and discontinuations. Where possible, reasons for change in treatment. Line of treatment.
Number of participant receiving supportive therapies while receiving palbociclib combination treatment | From 01 January 2015 to 30 September 2019
  Supportive therapies received since metastatic/locally advanced HR+/HER2- diagnosis while receiving palbociclib combination treatments. Duration of treatments.
Proportion of patients who are progression free at multiple intervals | From date of index treatment to date of disease progression, date of death, or end of study whichever came first, assessed up to 57 months
  Proportion of progression free survival/time to progression (at intervals per standard of care) (eg. 12, 18 months).
Objective response rate (ORR) | From date of index treatment up to 57 months
  Proportion of objective response rate (at intervals per standard of care).
Proportion of patients alive 1 and 2 years post palbociclib combination initiation depending on availability of follow-up data (if available) | From 01 January 2015 to 30 September 2019

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer; Meteb Al-Foheidi, Principal Investigator — King Abdul-Aziz Medical City, National Guard Hospital
Locations (7):
- Hamad Medical Corporation, Doha, Qatar
- Saudi Arabia (3):
  - King Abdulaziz Medical City National Guard Hospital, Jeddah
  - King Abdulaziz Medical City National Guard Hospital Riyahd, Riyadh
  - King Saud University Medical City Riyadh PO BOX 7805, Riyadh
- United Arab Emirates (3):
  - Tawam, Al Ain City
  - Dubai Hospital, Dubai
  - Mediclinic City Hospital, Dubai

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A5481136